CLINICAL TRIAL: NCT06001216
Title: The Relationship of Acute-Chronic Workload Ratio and Functional Movement Screen With Injury Risk in Adolescent Team Sport Players
Brief Title: The Relationship of ACWR and FMS With Injury Risk in Adolescent Players
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Aynur Demirel, Associate Professor, Hacettepe University
Other Study IDs: GO 21/1377
Record Dates: First submitted 2023-08-14; First posted 2023-08-21 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Injury;Sports
MeSH Terms: conditions — Athletic Injuries

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In this study, we examine how acute to chronic workload ratio and functional movement screen scores relate to injury risk in teenage athletes who play team sports.

DETAILED DESCRIPTION:
At least 60 volunteer athletes who have played team sport for at least 1 year, have not been away from the field for more than 2 weeks, 15 years and older are planned to include this study. All participating athletes in this study will sign an informed consent form then their demographic information will be recorded. The injury risk of athletes will be evaluated by functional movement screen. The functional movement screen is a test battery consisting of 7 tests. These tests are deep squat, hurdle step, in-line lunge, active straight-leg raise, trunk stability push-up, rotary stability and shoulder mobility. To calculate the acute-chronic workload, internal workloads during training and/or matches will be added up over a period of 8 weeks. As part of the study, health professionals on the team will provide injury information for the athletes. Sports injuries will be classified based on the type of injury (contact or non-contact) and the area of the body affected. The severity of the injury will be determined as follows: minimal (1-3 days of missed sports activity), mild (4-7 days of missed sports activity), moderate (1-4 weeks of missed sports activity), and severe (4 or more weeks of missed sports activity).

ELIGIBILITY:
Inclusion Criteria:

* Be over 16 years old,
* Participating in a team sport for at least one year,
* The players who have not stayed away from their sport for more than two weeks,

Exclusion Criteria:

* Any history of orthopedic or neurological injury or pain that may interfere with normal training or competition during assessment,
* Structural deformities such as scoliosis and leg length inequality,
* Their level of activity differs from other athletes in the same sport will be excluded from the study.

Ages: 15 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: All volunteer employees who are over the age of 15, have been playing a team sport for at least one year, have not been away from their spor for more than two weeks and meet the inclusion criteria of the study will be included.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-08-18 (Estimated); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
Functional Movement Screen | baseline
  To assess the risk of injury, we will utilize the Functional Movement Screen.The FMS test scores range from 0 to 3, with 0 being the worst and 3 being the best. The highest possible score is 21. Individuals who score 14 points or lower are at a higher risk for injury, while those who score above 14 points have a lower risk of injury.
Acute chronic workload ratio | 8 weeks
  To determine an athlete's workload, we ask them to rate their training time and fatigue level using the modified Borg scale after each session. We then calculate the workload by dividing the acute workload by the chronic workload using specific formulas.
Injury | 8 weeks
  The input will be provided by the health professionals on the team.